CLINICAL TRIAL: NCT01616953
Title: Cell Therapy for Craniofacial Bone Defects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Darnell Kaigler, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00060042
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Results first posted 2017-05-04 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-03

CONDITIONS: Cleft Palate; Trauma
Keywords: dental implants
MeSH Terms: conditions — Cleft Palate; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ixmyelocel-T (Experimental): iliac bone marrow aspirates are expanded ex vivo to enrich for adult multipotent cells (ixmyelocel-T) capable of regenerating bone and blood vessels and reducing inflammation. Following cell expansion, autologous ixmyelocel-T is then packaged and can be used as an autologous graft for treatment of bone defects.
  Interventions: Biological: Ixmyelocel-T
- Autogenous Bone Grafting (Active Comparator): Alveolar grafting will be performed. Under local anesthesia, and possibly conscious intravenous sedation (depending on patient desire for sedation due to anxiety), alveolar grafting will be performed with an autogenous bone block harvested from an intraoral or extraoral site, according to standard of care.
  Interventions: Procedure: Autogenous Bone Grafting

INTERVENTIONS:
Biological: Ixmyelocel-T — Twelve days after the bone marrow aspiration, alveolar grafting will be performed. Under local anesthesia, and possibly conscious intravenous sedation (depending on patient desire for sedation due to anxiety), alveolar grafting will be performed with the cell therapy (Ixmyelocel-T)
  Other Names: bone repair cells
  Arms: Ixmyelocel-T
Procedure: Autogenous Bone Grafting — Alveolar grafting will be performed. Under local anesthesia, and possibly conscious intravenous sedation (depending on patient desire for sedation due to anxiety), alveolar grafting will be performed with an autogenous bone block harvested from an intraoral or extraoral site, according to standard of care.
  Arms: Autogenous Bone Grafting

SUMMARY:
The purpose of this research is to determine if a patient's own bone marrow tissue can help regenerate bone in the area of the jaw where an implant will be placed. The name of the process is called Bone Repair Cell (BRC) Therapy. A sample of bone marrow tissue will be collected and sent to a laboratory where it will be processed to form more cells. These new cells will then be transplanted in the regenerative site. The researchers are testing to see if these cells (BRC) will help form bone. The research will also determine if the implant will be more stable in the area with new bone growth.

DETAILED DESCRIPTION:
Up to 20 (twenty) subjects who have alveolar defects secondary to clefts (n=10) or trauma (n=10), will be selected to participate in this study. Among the 20 patients, a total of up to 60 defect sites will be evaluated for bone regeneration following therapy, with each subject being evaluated in from one to four sites. Once enrolled, subjects from each of the two groups (cleft or trauma) will be randomly assigned to receive one of two possible treatments, traditional autogenous bone grafting or cell therapy (ixmyelocel-T)

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18 to 60 yrs
* Gender: Male and female
* Patients must be able and willing to follow study procedures and instructions.
* Patients must have read, understood and signed an informed consent for
* Missing tooth criteria:

  * Patients missing at least one maxillary lateral incisor secondary to cleft lip and/or palate:

    * with compromised bone support for installation of dental implant(s) ( > 3 mm deficiency in horizontal and/or vertical bone height)
    * with adequate interdental arch space for dental implant restorations
    * with bony continuity between cleft segments
    * with adequate interproximal space (between adjacent teeth) for dental implant installation
  * Patients missing multiple (1-4 teeth) teeth secondary to trauma:

    * in maxillary or mandibular anterior segments (second premolar to second premolar)
    * with compromised bone support for installation of dental implant(s) ( > 3 mm deficiency in horizontal and/or vertical bone height)
    * with adequate interdental arch space for dental implant restorations

Exclusion Criteria:

* Allergies or hypersensitivities to study related medications: dexamethasone, chlorhexidine, ibuprofen. For patients allergic to amoxicillin a comparable substitute antibiotic will be used.
* Hematologic disorders/ blood dyscrasias. Patients will have blood drawn for a complete blood count (CBC) test. Current University of Michigan Health System normal lab values are as follows: white blood count (WBC: 4.0-10.0 x103/cmm), red blood count (RBC: male 4.50-5.90 x103/cmm; female 3.90-5.30x103/cmm), hemoglobin (HgB: male 13-17.3gm/dl; female 12-16gm/dl), Hct (male 39-50.2%; female 35-48%), mean corpuscular volume (MCV: 80-100fl), mean corpuscular hemoglobin (MCH: 25-35 pg), mean corpuscular hemoglobin concentration (MCHC: 30-37%), red cell distribution width (RDW: 11.5-15.5%), Plt (150-450x103/cmm).
* Active infectious disease
* Liver or kidney dysfunction/failure- Patients will have blood drawn for serum laboratory tests, including creatinine, blood urea nitrogen, aspartate aminotransferase test (AST), alanine aminotransferase test (ALT), and bilirubin.
* All of these must be within normal limits for a patient to be included in the study.
* Current University of Michigan Health System normal lab values are as follows: *Creatinine (male 0.7-1.3 mg/dl

  * female 0.5-1.0 mg/dl)
  * blood urea nitrogen (BUN: 8-20 mg/dl)
  * AST (8-30 IU/L)
  * ALT (7-35 IU/L)
  * Bilirubin (0.2-1.2 mg/dl).
* Laboratory values that will define normal renal and hepatic function, as well as criteria for exclusion of metabolic bone disease are consistent with those established by the University of Michigan Health System (UMHS).
* Normal clinical values will be used to help assure the health of all subjects in this trial.
* Potential subjects whose laboratory values fall outside the UMHS normal ranges will be required to have medical clearance from their primary care provider prior to participation.
* Endocrine disorders/dysfunctions (i.e uncontrolled Type I or II diabetes, glycosylated hemoglobin [HA1C > 7%})
* Cancer - The explicit definition of cancer used to exclude patients is consistent with that described by the National Cancer Institute (NCI), National Institutes of Health. According to NCI, cancer is any disease in which abnormal cells divide without control and invade nearby tissues (invasive disease). These include carcinomas, sarcomas, leukemias, and lymphomas. Any patient with a history of these invasive diseases will be excluded from the study.
* Patients who currently use bisphosphonates or have a history of bisphosphonate use will be excluded from the trial.
* HIV+
* Metabolic Bone Diseases- Patients with metabolic bone diseases such as Paget's disease, hypercalcemia, moderate to severe vitamin D3 abnormalities or any other metabolic bone disease including osteoporosis and osteoporotic fractures will be excluded. The following scale will be used to determine osteoporosis in patients who have had a bone mass density (BMD determination: Normal = T score at or above -1.0 standard deviation [SD]); Osteopenia = T score between -1.0 and -2.5 SD; Osteoporosis = T score at or below -2.5 SD.
* Pregnant women- Female patients who are of childbearing potential are excluded except those who are using hormonal or barrier methods of birth control (oral or parenteral contraceptives, diaphragm plus spermicide, or condoms). Pregnancy status will be determined with a urine test and patients who are pregnant, as determined by a positive test, will be excluded from the study
* Patients with congenital or metabolic bone disorders
* Subjects with co-morbid conditions that would affect the study outcome or interpretation of study results will be excluded
* Subjects on significant concomitant drug therapy for systemic conditions (i.e. cardiovascular disease, renal dysfunction) will not be included in the study. Occasional short term use (7-14 days) of analgesics or common cold medication is permitted. Such use of these medications will be reviewed and recorded by the Investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darnell Kaigler, DDS, PhD, Principal Investigator — University of Michigan
Locations (1):
- Michigan Center for Oral Health Research, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ixmyelocel-T | Autogenous Bone Grafting
Started | 10 | 8
Implant Placement Surgery | 9 | 8
Implant Uncovery | 8 | 8
6 Months Post-loading | 8 | 8
Completed | 8 | 8
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — lack of bone and soft tissue | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixmyelocel-T | Autogenous Bone Grafting | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 27 [18 to 42] | 31 [19 to 54] | 29 [18 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 18
Pre-operative alveolar bone width [Mean (Standard Deviation); unit: millimeters] — The alveolar crest width at baseline was measured with a vernier caliper to the nearest half of a millimeter, 3mm below the crest
  millimeters | 2.6 (1.6) | 5 (1.1) | 3.8 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Bone Regeneration
Description: The primary outcome variables for bone regeneration will be measured by histological and microcomputed tomographic (μCT) analyses at 4 months post-grafting.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: implant sites
Arm/Group | Ixmyelocel-T | Autogenous Bone Grafting
Number analyzed (Participants) | 9 | 8
implant sites | 1.5 (1.5) | 3.3 (1.4)

2. Secondary Outcome: Implant Stabilization
Description: The ability of the dental implant fixtures to be loaded and remain stable for six months following implant loading (at 4 months) will be evaluated.
Time Frame: 10 months
Measure: Number; unit: participants
Arm/Group | Ixmyelocel-T | Autogenous Bone Grafting
Number analyzed (Participants) | 10 | 8
participants | 5 | 8

ADVERSE EVENTS:
Time Frame: August 2012 - June 2015
Arm/Group | Ixmyelocel-T | Autogenous Bone Grafting
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/8
Other Adverse Events (participants affected / at risk) | 9/10 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixmyelocel-T (N=10) | Autogenous Bone Grafting (N=8)
Car accident (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixmyelocel-T (N=10) | Autogenous Bone Grafting (N=8)
Tooth sensitivity (General disorders) | 1 (1) | 0 (0)
Infection of surgical site (Infections and infestations) | 1 (1) | 0 (0)
Mucosal ulcers (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Non-study implant failing (Surgical and medical procedures) | 1 (1) | 0 (0)
Streptococcal pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Self diagnosed inflamed rotator cuff (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Early suture removal (General disorders) | 0 (0) | 1 (1) — Subject chewing on surgical site
Wisdom teeth impactions (General disorders) | 1 (1) | 0 (0)
Non-study implant in sinus (General disorders) | 1 (1) | 0 (0)
Inflammation of wrist (Infections and infestations) | 1 (1) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0)
Incision line opening (General disorders) | 3 (3) | 0 (0)
Skin rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Swelling (Infections and infestations) | 3 (3) | 0 (0)
Tooth fracture (unrelated to study) (General disorders) | 1 (1) | 0 (0)
Unrelated bone graft procedure (General disorders) | 0 (0) | 1 (1)
Root #9 extraction (General disorders) | 0 (0) | 1 (1)
Left knee pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Torn ligament in ankle (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (General disorders) | 1 (1) | 1 (1)
Pain in recipient site (General disorders) | 0 (0) | 1 (1)
Membrane exposure (General disorders) | 1 (1) | 0 (0)
Localized erythema (General disorders) | 1 (1) | 1 (1)
Pain and dysesthesia in donor site (General disorders) | 0 (0) | 1 (1)
Early implant failure (General disorders) | 0 (0) | 1 (1)
Abutment screw broke (General disorders) | 1 (1) | 0 (0)
Implant restoration came off (General disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes